CLINICAL TRIAL: NCT00204308
Title: Addition of Single-dose, Maternal Tenofovir and Emtricitabine to Reduce Non-nucleoside Reverse Transcriptase Inhibitor Resistance Mutations in the Setting of Zidovudine and Nevirapine for Prevention of Mother-to-child HIV Transmission
Brief Title: Maternal TDF and FTC to Reduce NNRTI Resistance Mutations After Intrapartum NVP
Acronym: TD-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Responsible Party: Principal Investigator, Benjamin Chi, MD, MSc, Associate Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EGSA 19-02
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: HIV; Pregnancy
Keywords: HIV; Pregnancy; Mother-to-child transmission of HIV; Drug resistance; Nevirapine resistance; NNRTI resistance
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- combination tenofovir-emtricitabine (Experimental)
  Interventions: Drug: Combination tenofovir-emtricitabine
- control arm (No Intervention)

INTERVENTIONS:
Drug: Combination tenofovir-emtricitabine — Tenofovir disoproxil 300 mg / emtricitabine 200 mg taken as a single dose during labor
  Other Names: Truvada
  Arms: combination tenofovir-emtricitabine

SUMMARY:
The purpose of this study is to determine whether the addition of tenofovir (TDF) and emtricitabine (FTC)to a standard PMTCT regimen containing single-dose nevirapine (NVP) can reduce the development of post-ingestion HIV resistance to non-nucleoside reverse transcriptase inhibitors (NNRTIs).

DETAILED DESCRIPTION:
Single-dose intrapartum and neonatal nevirapine (NVP), either alone or in combination with short course zidovudine (ZDV) is in widespread use to prevent mother-to-child HIV transmission throughout the developing world. Though the public health benefits cannot be overstated, widespread use of NVP in this fashion may come at a cost. Non-nucleoside reverse transcriptase inhibitor (NNRTI) resistance mutations are induced in at least 20% and probably a larger proportion of women exposed to NVP in this fashion. Addition of short-course ZDV does not appear to mitigate this effect substantially. The full implications of these NVP resistance mutations are yet unknown, though there is concern that they may result in reduced efficacy of the NVP or other NNRTIs in long-term, therapeutic regimens.

We are conducting a clinical trial of tenofovir (TDF) and emtricitabine (FTC), marketed as a fixed dose combination, Truvada ™, to reduce NNRTI-resistance post-delivery in the setting of NVP with or without ZDV for PMTCT. TDF and FTC are both Category B drugs and are approved for use in pregnancy. They have several characteristics that make them ideal candidate drugs for use in conjunction with NVP, including long intracellular half-lives and established safety profile among adults for HIV treatment.

Women will be enrolled between 28 and 38 weeks of gestation. As part of normal PMTCT services, they may choose NVP-boosted ZDV or single dose NVP for PMTCT; We anticipate that most (~80%) will choose the former. At arrival for delivery, they will be randomized to receive either the two study drugs (intervention) or no drug (control). A total of 400 women will be randomized, and followed, along with their infants, for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Serologically confirmed HIV infection;
* Gestational age of 28 to 38 weeks;
* Previous selection of a NVP-based PMTCT regimen (with or without ZDV)
* Willingness to participate in a randomized trial;
* Willingness to follow up in a postpartum visit schedule;
* Willingness to allow her infant to participate in this trial;

Exclusion Criteria:

* Use of antiretroviral medications before this pregnancy, even in a single dose.
* Current use of antiretroviral medications for treatment of advanced HIV disease and/or AIDS
* Illness or complication of pregnancy likely to warrant transfer to the University Teaching Hospital (UTH), known at time of randomization;
* Known or suspected allergy to NVP or other benzodiazepine medications;
* History of known liver disease.
* Hemoglobin level of 7.9 g/dL or less

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2005-03; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
maternal antiretroviral drug resistance to non-nucloeoside reverse transcriptase inhibitors | 6 weeks

SECONDARY OUTCOMES:
maternal antiretroviral drug resistance to non-nucloeoside reverse transcriptase inhibitors | 2 weeks
maternal hematological and renal function after TDF-FTC use | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S A Stringer, MD, Principal Investigator — University of Alabama at Birmingham; Benjamin H Chi, MD, Study Director — University of Alabama at Birmingham
Locations (2):
- Zambia (2):
  - Kalingalinga Health Centre, Lusaka
  - Kanyama Health Centre, Lusaka

REFERENCES:
- [Result] Chi BH, Sinkala M, Mbewe F, Cantrell RA, Kruse G, Chintu N, Aldrovandi GM, Stringer EM, Kankasa C, Safrit JT, Stringer JS. Single-dose tenofovir and emtricitabine for reduction of viral resistance to non-nucleoside reverse transcriptase inhibitor drugs in women given intrapartum nevirapine for perinatal HIV prevention: an open-label randomised trial. Lancet. 2007 Nov 17;370(9600):1698-705. doi: 10.1016/S0140-6736(07)61605-5. Epub 2007 Nov 7. PMID 17997151
- [Result] Chi BH, Chintu N, Cantrell RA, Kankasa C, Kruse G, Mbewe F, Sinkala M, Smith PJ, Stringer EM, Stringer JS. Addition of single-dose tenofovir and emtricitabine to intrapartum nevirapine to reduce perinatal HIV transmission. J Acquir Immune Defic Syndr. 2008 Jun 1;48(2):220-3. doi: 10.1097/QAI.0b013e3181743969. PMID 18520682
- [Result] Chi BH, Ellis GM, Chintu N, Cantrell RA, Sinkala M, Aldrovandi GM, Warrier R, Mbewe F, Nakamura K, Stringer EM, Frenkel LM, Stringer JS. Intrapartum tenofovir and emtricitabine reduces low-concentration drug resistance selected by single-dose nevirapine for perinatal HIV prevention. AIDS Res Hum Retroviruses. 2009 Nov;25(11):1099-106. doi: 10.1089/aid.2009.0088. PMID 19886836
- [Result] Dorton BJ, Mulindwa J, Li MS, Chintu NT, Chibwesha CJ, Mbewe F, Frenkel LM, Stringer JS, Chi BH. CD4+ cell count and risk for antiretroviral drug resistance among women using peripartum nevirapine for perinatal HIV prevention. BJOG. 2011 Mar;118(4):495-9. doi: 10.1111/j.1471-0528.2010.02835.x. Epub 2010 Dec 24. PMID 21199294